CLINICAL TRIAL: NCT00523302
Title: A Pilot Study of Transcranial Magnetic Stimulation (TMS) Effects on Pain and Depression in Patients With Fibromyalgia
Brief Title: A Pilot Study of TMS Effects on Pain and Depression in Patients With Fibromyalgia
Acronym: TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR#17365; AR049459 (Other Grant/Funding Number: Multidisciplinary Clinical Research Center Grant P60)
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-05

CONDITIONS: Major Depression; Fibromyalgia
Keywords: Major Depression; Fibromyalgia; TMS
MeSH Terms: conditions — Depressive Disorder, Major; Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active TMS (Active Comparator): Since cortical stimulation can be performed non-invasively by active Transcranial Magnetic Stimulation (TMS), Participants in the active TMS group, receive five 20 minute active TMS treatment sessions per week for two weeks.
  Interventions: Device: Active TMS
- Sham TMS (Sham Comparator): To prevent unwanted cortical activation, Sham TMS will be employed in the Sham TMS group. For the Sham TMS group, a specially designed sham TMS coil will be used for all sham conditions. This sham TMS coil produces auditory signals identical to active TMS coils but is shielded so that actual stimulation does not occur. This approach is currently the state-of-the-art approach to sham TMS procedures and is employed in high-quality clinical TMS trials. Participants in the sham TMS group receive five 20 minute Sham TMS treatment sessions per week for two weeks.
  Interventions: Device: Sham TMS

INTERVENTIONS:
Device: Active TMS — Active TMS uses the active TMS coil to stimulate the cortical area of interest. Active TMS involves 80 trains x 15 sec = 4000 pulses per session, 5 x per week= 20,000 pulses per week, x 2 weeks = 40,000 pulses.
  Other Names: Neotonus model 2100 xxx
  Arms: Active TMS
Device: Sham TMS — Sham TMS uses the same stimulation frequency as the Active TMS but uses the Sham TMS coil instead to prevent actual stimulation from occurring (chosen as a priori stimulation based on studies showing antidepressant and anti-nociceptive effects): 10 Hertz - Pulse train duration (on time) 5 seconds, Power (intensity) level 120% of stored motor threshold, Inter-train interval (off time) 10 seconds (15 second cycle time). Additionally, stimulation-train duration and inter-stimulus intervals were determined such that they are in compliance with current published rTMS safety guidelines.
  Other Names: Neotonus model 2100 xxx
  Arms: Sham TMS

SUMMARY:
In this pilot study, the PI proposes to include 20 African American participants with Fibromyalgia to explore the effect of r TMS on pain and depressive symptoms.

DETAILED DESCRIPTION:
In this pilot study, the PI proposes to include 20 African American participants with Fibromyalgia to explore the effect of r TMS on pain and depressive symptoms. The focus on African Americans is due to the mandate from the funding source (internal), as well as possible higher prevalence of FM in AA women. If recruitment is slow, the PI proposes to open up the study to other groups. Twenty subjects will be randomized to either sham or active TMS condition. Inclusion/exclusion criteria are well thought out and seem appropriate. mTreatments will be administered at IOP 5 times/wk with each session lasting 20 minutes. Pain intensity and unpleasantness will be measured pre and post each TMS session using three different pain evaluation paradigms. GCRC resource is mainly requested for two blood draws pre and post first TMS session. The blood samples will be used to measure inflammatory cytokines IL-1, IL-6, AND IL-8. The main aim is to ascertain feasibility of the study and secondary aim is to gather information on variability in response for power analysis for future larger study. The introduction and rationale (including pain evaluation, and methods relating to TMS) are clearly presented. Use of GCRC resources seem appropriate.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80,
* meet ACR criteria for FM for more than 6 months,
* may or may not have a diagnosis of major depressive disorder (not bipolar) past or present,
* Current major depressive episode must be without psychotic features
* Not be on medication known to increase risk of TMS-induced seizures
* No prescription medication changes in the previous 4 weeks with agreement not to change during the treatment course (2 weeks) and 2 weeks thereafter
* No history of epilepsy or stroke or recent head trauma (LOC > 5 minutes) within the past 6 months
* African Americans will be initially sought out for study, however the recruitment may extend to include Caucasian and Hispanic subjects to carry out the study.

Exclusion Criteria:

* Primary, current diagnosis of schizophrenia
* Other (non-mood disorder) psychosis
* Mental retardation
* Substance dependence or abuse within the past 6 months (except nicotine)
* Psychotic features in this episode, dementia, or delirium
* Contraindication to rTMS
* Increased intracranial pressure
* Brain surgery, or head trauma with loss of consciousness for > 15 minutes
* Implanted electronic device
* Metal in the head, or pregnant
* Has an active autoimmune, endocrine, viral, or vascular disorder affecting the brain or unstable cardiac disease
* Uncontrolled hypertension, or severe renal or liver insufficiency
* Unstable and active suicidal intent or plan
* History of attempt requiring medical hospitalization within in the past 6 months
* -currently an involuntary inpatient on a psychiatric ward.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Short, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Short BE, Borckardt JJ, Anderson BS, Frohman H, Beam W, Reeves ST, George MS. Ten sessions of adjunctive left prefrontal rTMS significantly reduces fibromyalgia pain: a randomized, controlled pilot study. Pain. 2011 Nov;152(11):2477-2484. doi: 10.1016/j.pain.2011.05.033. Epub 2011 Jul 20. PMID 21764215

RESULTS

PARTICIPANT FLOW:
Groups:
- Active TMS: Participants receive 5 Active TMS treatment sessions per week for two weeks. Active stimulation involves 80 trains x 15 sec = 4000 pulses per session, 5 x per week= 20,000 pulses per week, x 2 weeks = 40,000 pulses. Time - 1200 sec = 20 minutes/ session, all days.
  Active TMS: Active TMS involves 80 trains x 15 sec = 4000 pulses per session, 5 x per week= 20,000 pulses per week, x 2 weeks = 40,000 pulses. Time - 1200 sec = 20 minutes/ session, all days.
- Sham TMS: Participants receive 5 Sham TMS treatment sessions per week for two weeks. Sham stimulation involves 80 trains x 15 sec = 4000 pulses per session, 5 x per week=20,000 pulses per week, x 2 weeks = 40,000 pulses. Time - 1200 sec = 20 minutes/ session, all days.
  Sham TMS: Sham TMS will use the same stimulation frequency for all active subjects (chosen as a priori stimulation based on studies showing antidepressant and anti-nociceptive effects): 10 Hertz - Pulse train duration (on time) 5 seconds, Power (intensity) level 120% of stored motor threshold, Inter-train interval (off time) 10 seconds (15 second cycle time). Additionally, stimulation-train duration and inter-stimulus intervals were determined such that they are in compliance with current published rTMS safety guidelines.
Period: Overall Study
Arm/Group | Active TMS | Sham TMS
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TMS | Sham TMS | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.20 (8.28) | 51.67 (18.19) | 53 (13.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Average Pain
Description: To assess each participant's average Pain in the past 24 hours, The Brief Pain Inventory (BPI)-short form will be administered. The BPI rapidly assesses the severity of pain and its impact on functioning and has been widely used in both research and clinical settings. Participants rate their average pain in the past 24 hours using a 0-10 numerical rating scale, where 0=no pain and 10=extreme pain.
Time Frame: Baseline, After Week 1 of Treatment, After Week 2 of Treatment, One week Post Treatment follow up, and Two week post treatment follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active TMS: Since cortical stimulation can be performed non-invasively by active Transcranial Magnetic Stimulation (TMS), Participants in the active TMS group, receive five 20 minute active TMS treatment sessions per week for two weeks. Active TMS uses the active TMS coil to stimulate the cortical area of interest. Active TMS involves 80 trains x 15 sec = 4000 pulses per session, 5 x per week= 20,000 pulses per week, x 2 weeks = 40,000 pulses.
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 5.60 (1.85) | 5.43 (1.82)
  After Week 1 of Treatment | 4.90 (1.89) | 5.49 (1.90)
  After Week 2 of Treatment | 3.99 (1.90) | 5.07 (1.89)
  1 week post treatment follow up | 4.19 (1.90) | 4.76 (1.90)
  2 week post treatment follow up | 4.41 (1.95) | 5.37 (2.02)

2. Primary Outcome: THE FIBROMYALGIA IMPACT QUESTIONNAIRE (FIQ)-Modified
Description: To assess the impact of fibromyalgia on each participant's function, the FIQ-modified (2002) version will be administered before each study visit. The FIQ-modified (2002) version assesses the following symptoms; physical Impairment, well-being, pain, fatigue, rested, stiffness, anxiety, and depression within the past 24 hours. Each symptom scale ranges from 0 to 10. For example, 0=no pain and 10=extreme pain, 0=not fatigued and 10=extremely fatigued.
  The final score is the total score which ranges from 0 to 80. Higher scores indicate greater impact of fibromyalgia on functioning.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 58.79 (11.93) | 54.38 (13.96)
  After Week 1 of Treatment | 55.03 (16.93) | 51.22 (15.96)
  After Week 2 of Treatment | 42.07 (18.13) | 51.50 (17.32)
  1 week Post Treatment follow up | 49.29 (19.27) | 43.47 (16.10)
  2 week Post Treatment follow up | 38.99 (19.44) | 47.93 (14.70)

3. Primary Outcome: THE HAMILTON DEPRESSION RATING SCALE (HRDS)
Description: To assess each participant's level of depression, the HRDS will be administered. The HRDS is a 17-item clinician-rated scale that is designed to evaluate depressed mood, vegetative and cognitive symptoms of depression, and comorbid anxiety symptoms. Eight items are scored on a 5-point scale, ranging from 0-4, where 0=not present and 4=severe. Nine items are scored from 0-2, where 0=None, 1=Mild, and 2=Severe. The final, total score ranges from 0-52. Scores in the range of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression, and scores over 24 are indicative of severe depression.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 21.80 (7.79) | 17.60 (7.31)
  After Week 1 of Treatment | 17.30 (8.27) | 17.40 (8.42)
  After Week 2 of Treatment | 16.10 (8.19) | 15.30 (7.62)
  1 week post treatment follow up | 15.80 (8.74) | 17.20 (7.55)
  2 week post treatment follow up | 14.10 (9.42) | 16.40 (8.18)

ADVERSE EVENTS:
Time Frame: 5 Weeks
Arm/Group | Active TMS | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No